CLINICAL TRIAL: NCT01996423
Title: Impact of Vitamin D Supplementation on Clinical Severity and Immunologic Tolerance of Pediatric Atopic Dermatitis
Brief Title: Impact of Vitamin D Supplementation on Severity of Pediatric Atopic Dermatitis
Acronym: VIDATOPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-185; 1130615 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2013-11-11; First posted 2013-11-27 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; vitamin D
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplementation (Experimental): Subjects in the experimental arm will receive weekly vitamin D3 doses in oral suspension during 6 weeks. Weekly dose varies according to age group: VD3 8000 IU between ages 2-5.9 years, VD3 12000 IU between ages 6-11.9 years, VD3 16000 IU between ages 12-17.9 years.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive weekly placebo oral suspension during 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Other Names: Cholecalciferol
  Arms: Vitamin D3 supplementation
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oral vitamin D supplementation improves the clinical severity of atopic dermatitis in children. In addition, this study plans to evaluate the effects of vitamin D supplementation on several key aspects of the immune system of children with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis diagnosed according to Hanifin and Rajka criteria
* Age 2 - 17 years
* SCORAD 10 - 103

Exclusion Criteria:

* Active skin infection
* History of underlying illness causing immunosuppression within the past 2 years
* Immunosuppressors taken within the past month
* Parathyroid disease
* Sarcoidosis
* Acute or chronic renal disease
* Hyper or hypocalcemia
* Thyroid disease
* Osteomalacia or Paget's disease of bone
* Malabsorption
* Use of VD supplements (> 400 IU daily) or fish oil supplements in the past month
* Treatment for known VD deficiency in the last 6 months
* Treatment with moderate or high potency topical corticosteroids, oral or topical antibiotics, oral antivirals, immune enhancers, or topical calcineurin inhibitors in the past 7 days
* Phototherapy in the past month
* Autoimmune disease or immunodeficiency
* Planned trip to sunny climate during the 6-week study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in SCORAD index | baseline and 6 weeks
  Change in Scoring Atopic Dermatitis (SCORAD) index after 6 weeks of vitamin D3 (VD3) supplementation or placebo in children with atopic dermatitis.

SECONDARY OUTCOMES:
Changes in Th2 immunity | baseline and 6 weeks
  Eosinophil blood counts, serum IgE, Th2 lymphocytes among stimulated PBMCs, serum CCL17, CCL22, and CCL27.
Change in dendritic cell-mediated tolerance and regulatory T cells | baseline and 6 weeks
  Number and phenotype of blood dendritic cells and number of regulatory T cells.
Effect of VD3 supplementation on immunity to Staphylococcus aureus | baseline and 6 weeks
  Serum cathelicidin levels, S. aureus skin carriage, and specific IgE to staphylococcal enterotoxins.
Vitamin D receptor single nucleotide polymorphisms | baseline and 6 weeks
  Effect of VDR SNPs on the VD3 response.
Change in epidermal protein expression | 6 weeks
  Gene expression of epidermal proteins by PCR obtained from lesional and non-lesional tape stripping samples.

OTHER OUTCOMES:
Number of participants with adverse events | 6 weeks
  Adverse events of atopic dermatitis patients with VD3 and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Borzutzky, M.D., Principal Investigator — School of Medicine, Pontificia Universidad Católica de Chile; Carlos A Camargo Jr., M.D., DrPH, Study Director — Massachusetts General Hospital, Harvard University, Boston, USA; Cristian Vera, M.D., Study Director — School of Medicine, Pontificia Universidad Católica de Chile; Lorena Cifuentes, M.D., Study Director — School of Medicine, Pontificia Universidad Católica de Chile; Sergio Silva, M.D., Study Director — School of Medicine, Pontificia Universidad Católica de Chile
Locations (1):
- School of Medicine, Pontificia Universidad Católica de Chile, Santiago, Chile

REFERENCES:
- [Derived] Borzutzky A, Iturriaga C, Perez-Mateluna G, Cristi F, Cifuentes L, Silva-Valenzuela S, Vera-Kellet C, Cabalin C, Hoyos-Bachiloglu R, Navarrete-Dechent C, Cossio ML, Le Roy C, Camargo CA Jr. Effect of weekly vitamin D supplementation on the severity of atopic dermatitis and type 2 immunity biomarkers in children: A randomized controlled trial. J Eur Acad Dermatol Venereol. 2024 Sep;38(9):1760-1768. doi: 10.1111/jdv.19959. Epub 2024 Mar 14. PMID 38483248